CLINICAL TRIAL: NCT06738043
Title: Dexmedetomidine Infusion Versus Low Dose Ketamine Infusion as an Adjuvant in Bariatric Surgery: A Randomized Controlled Comparative Study
Brief Title: Dexmedetomidine Versus Ketamine as Adjuvants in Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla Shalaby, Anesthesiology, Intensive Care and Pain Management Resident, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/2024ANET15
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Postoperative Pain; Bariatric Surgery
Keywords: Dexmedetomidine; Ketamine; Opioid-Sparing Analgesia; Randomized Controlled Trial; Pain Management
MeSH Terms: conditions — Obesity; Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into three parallel groups: dexmedetomidine, ketamine, or control (placebo) groups, each receiving specific interventions based on the protocol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation will be concealed using sequentially numbered, sealed envelopes. A nurse not involved in patient care will open the envelope after induction of anesthesia to assign patients to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine Group (Experimental): Participants in this group will receive a bolus dose of dexmedetomidine (0.5 µg/kg ideal body weight) diluted in 0.9% normal saline over 10 minutes before induction of anesthesia. This will be followed by a continuous infusion of dexmedetomidine at 0.5 µg/kg/h until 10 minutes before the end of surgery.
  Interventions: Drug: Dexmedetomidine infusion
- Ketamine Group (Experimental): Participants in this group will receive a bolus dose of ketamine (0.3 mg/kg ideal body weight) diluted in 0.9% normal saline over 10 minutes before induction of anesthesia. This will be followed by a continuous infusion of ketamine at 0.3 mg/kg/h until 10 minutes before the end of surgery.
  Interventions: Drug: Ketamine infusion
- Control Group (Placebo Comparator): Participants in this group will receive a bolus dose of 0.9% normal saline over 10 minutes before induction of anesthesia. This will be followed by a continuous infusion of 0.9% normal saline until 10 minutes before the end of surgery.
  Interventions: Drug: Normal Saline Infusion (Placebo)

INTERVENTIONS:
Drug: Dexmedetomidine infusion — A bolus dose of dexmedetomidine (0.5 µg/kg ideal body weight) diluted in 0.9% normal saline is infused over 10 minutes before induction of anesthesia, followed by a continuous infusion at 0.5 µg/kg/h until 10 minutes before the end of surgery.
  Arms: Dexmedetomidine Group
Drug: Ketamine infusion — A bolus dose of ketamine (0.3 mg/kg ideal body weight) diluted in 0.9% normal saline is infused over 10 minutes before induction of anesthesia, followed by a continuous infusion at 0.3 mg/kg/h until 10 minutes before the end of surgery.
  Arms: Ketamine Group
Drug: Normal Saline Infusion (Placebo) — A bolus dose of 0.9% normal saline is infused over 10 minutes before induction of anesthesia, followed by a continuous infusion of 0.9% normal saline until 10 minutes before the end of surgery.
  Arms: Control Group

SUMMARY:
This randomized controlled trial aims to compare the analgesic efficacy of dexmedetomidine infusion versus low-dose ketamine infusion as adjuvants in bariatric surgery. The study includes 90 patients undergoing bariatric surgery at Menoufia University Hospital, randomized into three groups: dexmedetomidine, ketamine, and control (placebo). Primary outcomes include total morphine consumption intra- and post-operatively. Secondary outcomes include postoperative pain scores, total analgesic consumption, time to first analgesic request, hemodynamic parameters, and patient satisfaction. This study seeks to explore safer, more effective pain management strategies to minimize opioid use in bariatric surgery patients.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled interventional trial evaluating the analgesic efficacy and opioid-sparing effects of dexmedetomidine and low-dose ketamine as adjuvants in bariatric surgery. Ninety patients meeting the inclusion criteria will be enrolled and randomized into three groups:

* Dexmedetomidine Group: Patients will receive a bolus dose of dexmedetomidine (0.5 µg/kg) followed by a continuous infusion (0.5 µg/kg/h) until 10 minutes before the end of surgery.
* Ketamine Group: Patients will receive a bolus dose of ketamine (0.3 mg/kg) followed by a continuous infusion (0.3 mg/kg/h) until 10 minutes before the end of surgery.
* Control Group: Patients will receive an equal volume of normal saline as a placebo.

Objectives

The primary objective is to compare intra- and postoperative morphine consumption between groups. Secondary objectives include:

* Pain assessment using the Numeric Rating Scale (NRS) at multiple time points postoperatively.
* Time to first request for rescue analgesia.
* Hemodynamic stability (heart rate and mean arterial pressure).
* Patient satisfaction assessed using a 5-point scale.
* Incidence of adverse effects such as nausea, vomiting, bradycardia, and respiratory depression.

Study Protocol All patients will undergo standard preoperative assessments, including history, physical examination, and laboratory investigations. General anesthesia will be induced and maintained per institutional protocols. Postoperatively, pain management will follow a stepwise approach, with intravenous paracetamol as rescue analgesia.

Significance Given the high prevalence of obesity-related comorbidities, bariatric surgery patients are at increased risk for postoperative complications, particularly with opioid use. This study addresses the need for opioid-sparing pain management strategies, potentially reducing the risks of opioid-related adverse effects and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years.
* Both sexes.
* Body mass index (BMI) > 35 kg/m², scheduled for bariatric surgery.
* American Society of Anesthesiologists (ASA) physical status I-II.

Exclusion Criteria:

* History of hypersensitivity to dexmedetomidine or ketamine.
* History of substance abuse or chronic opioid use.
* American Society of Anesthesiologists (ASA) physical status III or IV.
* Severe hepatic or renal impairment.
* Cardiopulmonary disorders.
* Severe diabetes mellitus.
* Psychiatric disorders, seizures, uncontrolled hypertension (systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg), or heart block.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Total Morphine Consumption Intra- and Postoperatively | From the start of anesthesia to 24 hours postoperatively
  The total dose of morphine (measured in mg) consumed by participants intraoperatively and within the first 24 hours postoperatively. This includes morphine administered as part of the anesthesia protocol and as rescue analgesia post-surgery.

SECONDARY OUTCOMES:
Postoperative Pain Scores (Numeric Rating Scale - NRS) | At 1, 2, 4, 8, 12, 16, and 24 hours postoperatively
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain). Pain scores will be recorded at specific intervals postoperatively (1, 2, 4, 8, 12, 16, and 24 hours).
Time to First Request for Rescue Analgesia | 24 hours postoperatively
  The duration (in hours) from the end of surgery to the first request for rescue analgesia (intravenous morphine) by the participant.
Hemodynamic Stability (Heart Rate) | From baseline (pre-surgery) to 24 hours postoperatively
  Heart rate (HR) will be monitored and recorded at specific intervals during and after surgery to assess hemodynamic stability.
Hemodynamic Stability (Mean Arterial Pressure) | From baseline (pre-surgery) to 24 hours postoperatively
  Mean arterial pressure (MAP) will be monitored and recorded at specific intervals during and after surgery to assess hemodynamic stability.
Total Analgesic Consumption (Other Than Morphine) | At 24 hours postoperatively
  The total dose of non-morphine analgesics (e.g., paracetamol) administered postoperatively to manage pain within the first 24 hours after surgery.
Patient Satisfaction with Pain Management | At 24 hours postoperatively
  Patient satisfaction will be assessed using a 5-point Likert scale (1 = highly satisfied, 2 = satisfied, 3 = neutral, 4 = unsatisfied, 5 = highly unsatisfied) based on their postoperative pain management experience.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting information will be available starting 6 months after publication of the study results and will remain accessible for 5 years.
Access Criteria: Access to IPD and supporting information will be provided to qualified researchers upon reasonable request. Requests should include a proposal outlining the intended research objectives, ethical approval, and a data-sharing agreement. Access will be granted via secure data transfer or repository.